CLINICAL TRIAL: NCT04219397
Title: Investigating the Impact of Formal Interventions on Reducing Residual Opioids in the Home Following Legitimate Prescribing for Acute Post-surgical Pain in Pediatric Patients.
Brief Title: Investigating Interventions to Reduce Residual Opioids in the Home Following Legitimate Opioid Prescribing in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: The Society for Pediatric Anesthesia (Other); LCMC Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1905175369
Record Dates: First submitted 2019-12-13; First posted 2020-01-07 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Opioid Use, Unspecified
Keywords: opioid stewardship

STUDY DESIGN:
Intervention Model Description: 1. Usual care (control)
  2. Intervention #1: provision of formal education on medication take back
  3. Intervention #2: provision of formal education on medication home disposal of residual opioids, and provision of a medication home disposal kit.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Following patient enrollment, only the unblinded study coordinators will provide information and education to the patients/families about which arm they are randomized to. The investigator and other collaborators will conduct follow-up phone calls and data input and analysis in a blinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients in this group will receive usual care from the acute pain medicine service, and will go home with standardized multimodal analgesic protocol. There will be no interventions provided. They will receive a follow up phone call survey and be asked to return a completed medication education calendar that is provided as a part of usual APS care.
- Medication take back education intervention (Experimental): Patients in this group will receive usual care from the acute pain medicine service, and will go home with standardized multimodal analgesic protocol as described in the control group. They will receive a standardized education intervention. This intervention will educate patients and their families about medication take back programs, and will provide tailored directions to the closest medication take back center from their home, and also an option for medication take back that is located in close proximity to Riley Hospital clinics.
  Interventions: Other: Medication take back
- Home disposal kit intervention (Experimental): Patients in this group will receive usual care from the acute pain medicine service, and will go home with standardized multimodal analgesic protocol as described in the control group. They will receive standardized education about how to use the medication home disposal kit : Dispose Rx(r), and they will be instructed to use this kit to dispose of any left over opioid medications that they may have after they have competed therapy for pain management at home.
  Interventions: Other: Medication home disposal

INTERVENTIONS:
Other: Medication take back — Patients will be provided with formal education about medication take back programs for left-over prescription medications. They will be provided with directions to the closest medication take back facility to their home, and directions to the closet medication take back facility near their post-operative clinic site, and instructed to dispose of any left-over oxycodone medication (at completion of analgesic therapy) through participating in medication take back.
  Arms: Medication take back education intervention
Other: Medication home disposal — Patients and their families will be provided with formal education about how to use the medication home disposal kit: Dispose Rx, provided with a Dispose Rx home disposal kit, and instructed to dispose of any left-over oxycodone prescription medications with this kit following completion of analgesic therapy.
  Arms: Home disposal kit intervention

SUMMARY:
The overall objective of this study is to evaluate strategies to reduce unused opioids prescribed for pediatric acute post-surgical pain management.

DETAILED DESCRIPTION:
Prescription opioids are abused by an estimated 12.5 million Americans, and accidental opioid overdose is the leading cause of injury death in the US. Many of these drugs originate from leftover prescription opioids related to postoperative overprescribing, lack of proper disposal, and unsafe home storage. Governmental guidelines indicate that leftover prescription opioids should be preferentially returned to a drug take back site; however, many people do not utilize these programs due to travel distance, lack of transportation, or other factors.

The aims are to quantify the amount of unused opioids in the home following painful pediatric surgical procedures, investigate the impact of formal interventions on disposal of residual opioids in the home following these surgeries, and to identify current behaviors of adolescents and their family members in the handling of unused prescribed opioids.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children ages 12-17.9 years old
* ASA physical status 1 and 2
* Patients undergoing primary posterior spinal fusion surgery for correction of idiopathic scoliosis.
* Patients undergoing Nuss bar correction of pectus excavatum deformity.

Exclusion Criteria:

* Oxycodone allergy
* severe sleep apnea
* developmental delay
* neurological disorders
* liver disease/impairment
* renal disease/decreased renal function
* patients on opioid therapy prior to surgery
* Requires a translator for communication in English

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Quantification of residual opioids. | Post-discharge days 8-10
  Identify if there are left over opioid medications following completion of analgesic therapy, and if so, how many?
Assess participation in medication take back through follow up phone interview questionnaire. | Post-discharge days 8-10
  Assess the degree of participation in medication take back programs to dispose of any residual opioid medications following completion of analgesic therapy.
Assess participation in medication home disposal through follow up phone interview questionnaire. | Post-discharge days 8-10
  Assess the degree of participation in medication home disposal to dispose of any residual opioid medications following completion of analgesic therapy.

SECONDARY OUTCOMES:
Identify noncompliance/unsafe behaviors that contribute to retention of residual opioids through follow up phone interview questionnaire. | Post-discharge days 8-10
  Identify noncompliance/unsafe behaviors that contribute to retention of residual opioids despite formal education to patients/families about medication take back and medication home disposal of residual medications at the completion of analgesic therapy.
Average daily pain scores reported as values on Numerical Rating Scale. | Preoperatively through post-discharge day #10
  Assess average daily pain scores for patients undergoing painful surgeries in the perioperative period and following discharge from the hospital. This will be obtained through numerical report on study specific calendar. Numerical values are reported as a minimum of zero and a maximum of 10 on the Numerical Rating Scale. 0 corresponds with no pain, 1 with lower pain, and 10 corresponds with the most severe pain.
Frequency of opioid consumption through follow up phone interview questionnaire. | Post-operative day 1 through post-discharge day 10
  Assess the frequency of daily oxycodone consumption and correlate consumption with self reported pain scores. This measure will ask for a self-reported numerical frequency of daily opioid medication use. When this medication is used, we ask patients to rate their pain on the Numerical rating Scale from 0 to 10. Zero corresponds with no pain, 10 corresponds with the most severe pain.

OTHER OUTCOMES:
Demographic data | preoperatively through post-discharge day 10
  Obtain demographic data for study participants including: age, sex, race, ethnicity, and zip code as a marker of socioeconomic status, household income levels
Post operative pain scores reported as a numerical value on the Numerical Rating Scale. | Post operative day zero through post-discharge day 10
  Obtain post operative pain scores from post operative day zero through post discharge day 10. Pain scores are obtained as a numerical value on the Numerical Rating Scale. A score of zero corresponds with no pain, 1 is low pain, and 10 is the most severe pain.
Opioid consumption | Preoperatively through post-discharge day 10
  Assess total daily morphine equivalents
Prescription fill | Post discharge day 10
  Assess if the patient's prescription for oxycodone was filled
Actions related to residual opioids | Post discharge day 10
  Obtain qualitative information regarding the patient/families' intentions for what to do with left over opioid medications if they exist
Motivations for disposal of residual opioids obtained through study specific follow up phone call questionnaire. | Post discharge day 10
  Assess patient/family motivations for disposal of any residual opioids following completion of analgesic therapy.
Motivations for retention of residual opioids through study specific follow up phone interview questionnaire. | Post discharge day 10
  Assess patient/family motivations for retention of any residual opioids following completion of analgesic therapy
Barriers to disposal of residual opioids through study specific follow up phone interview questionnaire. | Post discharge day 10
  Assess patient/family barriers, if any, to disposal of residual opioids following completion of analgesic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michele A Hendrickson, MD,MS, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Riley Hospital for Children/Indiana University, Indianapolis, Indiana
  - Children's Hospital of New Orleans/ LCMC Health, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No